CLINICAL TRIAL: NCT02440321
Title: The Third Year Project of The Associated Factors of Smoking Around School-aged Children and The Intervention Development Using the Theory of Reasoned Action
Brief Title: Effects of Parent-child Interactive Intervention in Preventing Children's Environmental Tobacco Smoke Exposure at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, ping-ling Chen, Professor, Graduate Institute of Injury Prevention and Control, College of Public Health and Nutrition, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NSC97-2314-B-038-043-MY3
Record Dates: First submitted 2015-04-23; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Environmental Tobacco Smoke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- parent-child interactive program (Experimental): The parent-child interactive program is designed by three phase: precontemplation/ contemplation stage, preparation stage, and action/maintenance stage. In phase 1, the main focus is to promote motivation through information providing and being aware of children's perception toward ETS and smoking. In phase 2, the main focus is strengthening parents/children's ability to plan and implement smoke-free home. In phase 3, intervention focus is on maintaining behavioral change and smoke-free home by continuously strengthening implementing ability, identifying and eliminating barriers, and reinforcing successful experience. Parent-child interaction is designed through three phases, and parents perceive children's feedback through all phases.
  Interventions: Behavioral: Parent-child interactive program
- written materials (Active Comparator): The mailed materials included information on ETS and its adverse effects, smoking behavior that causes ETS at home, and a workbook for smoking cessation.
  Interventions: Other: written materials

INTERVENTIONS:
Behavioral: Parent-child interactive program
  Arms: parent-child interactive program
Other: written materials
  Arms: written materials

SUMMARY:
The purpose of this project is to develop and examine the effects of a parent-child interactive program to decrease the level of children's exposure to environmental tobacco smoke(ETS) at home, promote parents' and children's preventing strategy, knowledge of its hazard and attitude against environment tobacco smoke. A clustered randomized controlled trial was administered to school-aged children and their parents. The outcome indicators, children's exposure to ETS at home and increase of strategy to prevent the exposure were measured at baseline, 8 weeks, and 20 weeks. The other outcomes, parents' and children's knowledge of and attitude toward ETS, family's anti-ETS climate and its influence, and children's self efficacy of avoiding ETS were also measured at the same time point.

DETAILED DESCRIPTION:
Children exposing to environmental tobacco smoke (ETS) has been a global concern in public health. Home environment, especially parental smoking, has been identified as the major exposing source for children. Therefore parents' involvement becomes critical in preventing program. The purpose of this project is to develop and examine the effects of a parent-child interactive program to decrease the level of children's exposure to environmental tobacco smoke at home, promote parents' and children's preventing strategy, knowledge of its hazard and attitude against environment tobacco smoke. The other purposes included promoting family's anti-ETS climate that parents perceived and children's self-efficacy of ETS avoidant behavior.

A clustered randomized controlled trial was administered to 75 parents of school-aged children (ITT) and their children (parent-child dyads) from six primary schools in New Taipei City, Taiwan. Parent-child dyads in intervention group received a parent-child interactive program comprising three weekly group sessions and one individual telephone counseling session, which was administered 4 weeks after the group sessions. The participants in the control group received written materials related to tobacco information by mail four times during the same time period in place of the intervention sessions. The parent-child interactive intervention was developed according to the Transtheoretical Model and I-change Model. The main focuses of the intervention are to instill knowledge regarding the mechanism of the harmful effect of ETS, correct people's perceptions of the smoking patterns that lead to ETS exposure at home and effective and ineffective strategies for reducing ETS, and assist parent-child dyads in formulating strategies for maintaining a smoke-free home. The written materials mailed to participants in control group included information on ETS and its adverse effects, smoking behavior that causes ETS at home, and smoking cessation.

The outcome indicators were measured at baseline, 8 weeks, and 20 weeks. The primary outcome include children's exposure of ETS at home and prevention of children's ETS exposure. Children's exposure of ETS at home was measured by parents smoking at home and at the presence of the children for the last 7 days, and children's urinary cotinine level. The final collection of children's urine was performed 6 months after the intervention rather than 3 months after the intervention because of a delay in receiving urine cotinine measurement kits. Prevention of ETS exposure was measured by Parent-reported preventing strategies and child-reported avoiding behaviors. The second outcomes include parent/children reported knowledge of and attitude toward ETS, parents-reported family's anti-ETS climate and its influence, and children-reported their self-efficacy in avoiding ETS exposure. Collected data was analyzed by Chi-square test and generalized estimating equation. A pre-and-posttest pilot study on 10 parent-child dyads from two primary schools was conducted before this study.

ELIGIBILITY:
Inclusion Criteria:

* For parents：1. current smokers (people who smoked more than 100 cigarettes during their lifetime and had smoked within 30 days); 2. smoked at home over the past 7 days
* For children：the third to sixth grades of primary school

Exclusion Criteria:

* Children who had renal disease or were cognitively impaired according to their school teachers were excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change of Children's exposure of environmental tobacco smoke at home as measured by children's urine cotinine level, and questionnaire of parents smoking at home and in the presence of children for the last 7 days reported by parents and their children. | baseline, 8 week and 20 weeks for questionnaire/6 months for children's urine cotinine level.
  This outcome measure is a composite outcome consisting of bio-marker (cotinine) and self-reported data. Questions of parents smoking at home and in the presence of children for the last 7 days reported by parents and their children were modified from related items in the Adult Smoking Behavior Survey and Chinese Version of the Global Youth Tobacco Survey.
Parent reports Change of strategies for preventing children's exposure to environmental tobacco smoke at home as measured by developed questionnaire. | baseline, 8 weeks, and 20weeks
  The questionnaire was developed on the basis of a qualitative study and tested for content validity by 6 experts and internal consistency by using a sample of 182 parental smokers and their school-aged children who lived together. The mean item content validity index (CVI) for the entire scale was calculated resulting in a mean item CVI of 0.97. Cronbach's alpha for the scale was 0.72 in a prior survey of 182 parental smokers.
Child report change of environmental tobacco smoke avoidance behavior at home as measured by developed questionnaire. | baseline, 8 weeks, and 20weeks
  The questionnaire was based on the Avoidance of ETS scale originally developed by Martinelli and then translated and revised by Li and Wang. The CVI was 0.96, Cronbach's alpha for the scale was 0.89 in a previous study of 182 children of parental smokers.

SECONDARY OUTCOMES:
Parent and children reports change of knowledge of environment tobacco smoke hazard and attitude against environment tobacco smoke, as measured by developed questionnaires. | baseline, 8 weeks, and 20weeks
  The questionnaires were developed on the basis of a qualitative study and tested for content validity by 6 experts and internal consistency by using a sample of 182 parental smokers and their school-aged children who lived together. The mean item content validity index (CVI) was 0.87 to 0.97. Cronbach's alpha/KR 20 for the scale was 0.72 to 0.89 in a prior survey of 182 parental smokers and children.
Parent reports change of family's anti-smoking responses and parent's reaction to family's anti-smoking responses, as measured by developed questionnaires. | baseline, 8 weeks, and 20weeks
  The questionnaire was developed on the basis of a qualitative study and tested for content validity by 6 experts and internal consistency by using a sample of 182 parental smokers and their school-aged children who lived together. The mean item content validity index (CVI) was 0.94 to 0.97. Cronbach's alpha for the scale was 0.86 to 0.93 in a prior survey of 182 parental smokers.
change of children's self-efficacy in avoiding environmental tobacco smoke exposure, as measured by developed questionnaires. | baseline, 8 weeks, and 20weeks
  The questionnaire was based on the Self-efficacy of Avoiding ETS scale originally developed by Martinelli and then translated and revised by Li and Wang. The CVI was 0.94, Cronbach's alpha for the scale was 0.83 in a previous study of 182 children of parental smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Ling Chen, Ph.D., Principal Investigator — Graduate Institute of Injury Prevention and Control, College of Public Health and Nutrition, Taipei Medical University

REFERENCES:
- [Background] Craig, L., & Sawrikar, P. (2009). Work and Family: How Does the (Gender) Balance Change as Children Grow? Gender, Work & Organization, 16(6), 684-709. doi: 10.1111/j.1468-0432.2009.00481.x
- [Background] Grigsby, J. (1997). Telemedicine in the United States. In R. L. Bashshur, J. H. Sanders & G. W. Shannon (Eds.), Telemedicine: Theory and Practice (pp. 265-290). Springfield, IL: Charles C Thomas.
- [Background] Matt GE, Bernert JT, Hovell MF. Measuring secondhand smoke exposure in children: an ecological measurement approach. J Pediatr Psychol. 2008 Mar;33(2):156-75. doi: 10.1093/jpepsy/jsm123. Epub 2007 Dec 13. PMID 18079169
- [Background] Nierkens V, Stronks K, de Vries H. Attitudes, social influences and self-efficacy expectations across different motivational stages among immigrant smokers: replication of the O pattern. Prev Med. 2006 Oct;43(4):306-11. doi: 10.1016/j.ypmed.2006.05.005. Epub 2006 Aug 17. PMID 16919321
- [Background] Office on Smoking and Health (US). The Health Consequences of Involuntary Exposure to Tobacco Smoke: A Report of the Surgeon General. Atlanta (GA): Centers for Disease Control and Prevention (US); 2006. Available from http://www.ncbi.nlm.nih.gov/books/NBK44324/ PMID 20669524
- [Background] World Health Organization. (2009). Exposure to secondhand tobacco smoke and early death, at WHO Report on the Global Tobacco Epidemic, 2009: Implementing smoke-free environments
- [Result] Abdullah AS, Hitchman SC, Driezen P, Nargis N, Quah AC, Fong GT. Socioeconomic differences in exposure to tobacco smoke pollution (TSP) in Bangladeshi households with children: findings from the International Tobacco Control (ITC) Bangladesh Survey. Int J Environ Res Public Health. 2011 Mar;8(3):842-60. doi: 10.3390/ijerph8030842. Epub 2011 Mar 15. PMID 21556182
- [Result] Abdullah AS, Hua F, Xia X, Hurlburt S, Ng P, MacLeod W, Siegel M, Griffiths S, Zhang Z. Second-hand smoke exposure and household smoking bans in Chinese families: a qualitative study. Health Soc Care Community. 2012 Jul;20(4):356-64. doi: 10.1111/j.1365-2524.2011.01035.x. Epub 2011 Oct 27. PMID 22029412
- [Result] Abdullah AS, Mak YW, Loke AY, Lam TH. Smoking cessation intervention in parents of young children: a randomised controlled trial. Addiction. 2005 Nov;100(11):1731-40. doi: 10.1111/j.1360-0443.2005.01231.x. PMID 16277633
- [Result] Akhtar PC, Haw SJ, Currie DB, Zachary R, Currie CE. Smoking restrictions in the home and secondhand smoke exposure among primary schoolchildren before and after introduction of the Scottish smoke-free legislation. Tob Control. 2009 Oct;18(5):409-15. doi: 10.1136/tc.2009.030627. Epub 2009 Aug 10. PMID 19671536
- [Result] Aveyard P, Massey L, Parsons A, Manaseki S, Griffin C. The effect of Transtheoretical Model based interventions on smoking cessation. Soc Sci Med. 2009 Feb;68(3):397-403. doi: 10.1016/j.socscimed.2008.10.036. Epub 2008 Nov 27. PMID 19038483
- [Result] Baheiraei A, Kharaghani R, Mohsenifar A, Kazemnejad A, Alikhani S, Milani HS, Mota A, Hovell MF. Reduction of secondhand smoke exposure among healthy infants in Iran: randomized controlled trial. Nicotine Tob Res. 2011 Sep;13(9):840-7. doi: 10.1093/ntr/ntr085. Epub 2011 Apr 18. PMID 21504887
- [Result] Baldwin SA, Christian S, Berkeljon A, Shadish WR. The effects of family therapies for adolescent delinquency and substance abuse: a meta-analysis. J Marital Fam Ther. 2012 Jan;38(1):281-304. doi: 10.1111/j.1752-0606.2011.00248.x. Epub 2011 Sep 6. PMID 22283391
- [Result] Berman BA, Wong GC, Bastani R, Hoang T, Jones C, Goldstein DR, Bernert JT, Hammond KS, Tashkin D, Lewis MA. Household smoking behavior and ETS exposure among children with asthma in low-income, minority households. Addict Behav. 2003 Jan-Feb;28(1):111-28. doi: 10.1016/s0306-4603(01)00221-0. PMID 12507531
- [Result] Binnie V, McHugh S, Macpherson L, Borland B, Moir K, Malik K. The validation of self-reported smoking status by analysing cotinine levels in stimulated and unstimulated saliva, serum and urine. Oral Dis. 2004 Sep;10(5):287-93. doi: 10.1111/j.1601-0825.2004.01018.x. PMID 15315646
- [Result] Bolte G, Fromme H; GME Study Group. Socioeconomic determinants of children's environmental tobacco smoke exposure and family's home smoking policy. Eur J Public Health. 2009 Jan;19(1):52-8. doi: 10.1093/eurpub/ckn114. Epub 2008 Nov 25. PMID 19033356
- [Result] Bottorff JL, Oliffe J, Kalaw C, Carey J, Mroz L. Men's constructions of smoking in the context of women's tobacco reduction during pregnancy and postpartum. Soc Sci Med. 2006 Jun;62(12):3096-108. doi: 10.1016/j.socscimed.2005.11.058. Epub 2006 Jan 18. PMID 16414163
- [Result] Bureau of Health Promotion, D. o. H. (2010). Taiwan Tobacco Control Annual Report, 2010 Retrieved from http://tobacco.bhp.doh.gov.tw/Upload/FTB/UpFiles/2010.pdf
- [Result] Cahill K, Lancaster T, Green N. Stage-based interventions for smoking cessation. Cochrane Database Syst Rev. 2010 Nov 10;(11):CD004492. doi: 10.1002/14651858.CD004492.pub4. PMID 21069681
- [Result] Chan S, Lam TH. Protecting sick children from exposure to passive smoking through mothers' actions: a randomized controlled trial of a nursing intervention. J Adv Nurs. 2006 May;54(4):440-9. doi: 10.1111/j.1365-2648.2006.03842.x. PMID 16671973
- [Result] Chan SS, Lam TH, Salili F, Leung GM, Wong DC, Botelho RJ, Lo SL, Lau YL. A randomized controlled trial of an individualized motivational intervention on smoking cessation for parents of sick children: a pilot study. Appl Nurs Res. 2005 Aug;18(3):178-81. doi: 10.1016/j.apnr.2005.01.002. PMID 16106336
- [Result] Chen YT, Chung MC, Hsiao FH, Miao NF, Chen PL. Exploration of parental smokers' experience, perceptions, and family's influences on their smoking in the presence of children. ANS Adv Nurs Sci. 2012 Jan-Mar;35(1):E1-13. doi: 10.1097/ANS.0b013e3182445525. PMID 22293613
- [Result] Chen YH, Chen PL, Huang WG, Chiou HY, Hsu CY, Chao KY. Association between social climate for smoking and youth smoking behaviors in Taiwan: an ecological study. Int J Nurs Stud. 2010 Oct;47(10):1253-61. doi: 10.1016/j.ijnurstu.2010.02.007. Epub 2010 Mar 15. PMID 20233616
- [Result] Chen YT, Hsiao FH, Miao NF, Chen PL. Factors associated with parents’ perceptions of parental smoking in the presence of children and its consequences on children. Int J Environ Res Public Health. 2013 Jan 7;10(1):192-209. doi: 10.3390/ijerph10010192. PMID 23296207
- [Result] Conway TL, Woodruff SI, Edwards CC, Hovell MF, Klein J. Intervention to reduce environmental tobacco smoke exposure in Latino children: null effects on hair biomarkers and parent reports. Tob Control. 2004 Mar;13(1):90-2. doi: 10.1136/tc.2003.004440. PMID 14985605
- [Result] Curry SJ, Ludman EJ, Graham E, Stout J, Grothaus L, Lozano P. Pediatric-based smoking cessation intervention for low-income women: a randomized trial. Arch Pediatr Adolesc Med. 2003 Mar;157(3):295-302. doi: 10.1001/archpedi.157.3.295. PMID 12622686
- [Result] Dhar P. Measuring tobacco smoke exposure: quantifying nicotine/cotinine concentration in biological samples by colorimetry, chromatography and immunoassay methods. J Pharm Biomed Anal. 2004 Apr 1;35(1):155-68. doi: 10.1016/j.jpba.2004.01.009. PMID 15030890
- [Result] Dijk F, Reubsaet A, de Nooijer J, de Vries H. Smoking status and peer support as the main predictors of smoking cessation in adolescents from six European countries. Nicotine Tob Res. 2007 Sep;9 Suppl 3:S495-504. doi: 10.1080/14622200701587060. PMID 17978978
- [Result] Ding D, Wahlgren DR, Liles S, Jones JA, Hughes SC, Hovell MF. Secondhand smoke avoidance by preteens living with smokers: to leave or stay? Addict Behav. 2010 Nov;35(11):989-94. doi: 10.1016/j.addbeh.2010.06.016. Epub 2010 Jun 22. PMID 20634003
- [Result] Doubeni CA, Li W, Fouayzi H, Difranza JR. Perceived accessibility as a predictor of youth smoking. Ann Fam Med. 2008 Jul-Aug;6(4):323-30. doi: 10.1370/afm.841. PMID 18626032
- [Result] Ekerbicer HC, Celik M, Guler E, Davutoglu M, Kilinc M. Evaluating environmental tobacco smoke exposure in a group of Turkish primary school students and developing intervention methods for prevention. BMC Public Health. 2007 Aug 10;7:202. doi: 10.1186/1471-2458-7-202. PMID 17692111
- [Result] Emmons KM, Hammond SK, Fava JL, Velicer WF, Evans JL, Monroe AD. A randomized trial to reduce passive smoke exposure in low-income households with young children. Pediatrics. 2001 Jul;108(1):18-24. doi: 10.1542/peds.108.1.18. PMID 11433049
- [Result] Escoffery C, McCormick L, Bateman K. Development and process evaluation of a web-based smoking cessation program for college smokers: innovative tool for education. Patient Educ Couns. 2004 May;53(2):217-25. doi: 10.1016/S0738-3991(03)00163-0. PMID 15140462
- [Result] Farber HJ, Knowles SB, Brown NL, Caine L, Luna V, Qian Y, Lavori P, Wilson SR. Secondhand tobacco smoke in children with asthma: sources of and parental perceptions about exposure in children and parental readiness to change. Chest. 2008 Jun;133(6):1367-1374. doi: 10.1378/chest.07-2369. Epub 2008 Mar 13. PMID 18339788
- [Result] Fossum B, Arborelius E, Bremberg S. Evaluation of a counseling method for the prevention of child exposure to tobacco smoke: an example of client-centered communication. Prev Med. 2004 Mar;38(3):295-301. doi: 10.1016/j.ypmed.2003.10.008. PMID 14766111
- [Result] Green E, Courage C, Rushton L. Reducing domestic exposure to environmental tobacco smoke: a review of attitudes and behaviours. J R Soc Promot Health. 2003 Mar;123(1):46-51. doi: 10.1177/146642400312300115. PMID 12722583
- [Result] Gursoy ST, Soyer MT, Ocek Z, Ciceklioglu M, Aksu F. Why are Turkish children at risk of exposure to environmental tobacco smoke in their homes? Asian Pac J Cancer Prev. 2008 Jul-Sep;9(3):467-72. PMID 18990022
- [Result] Hannover W, Thyrian JR, Roske K, Grempler J, Rumpf HJ, John U, Hapke U. Smoking cessation and relapse prevention for postpartum women: results from a randomized controlled trial at 6, 12, 18 and 24 months. Addict Behav. 2009 Jan;34(1):1-8. doi: 10.1016/j.addbeh.2008.07.021. Epub 2008 Aug 3. PMID 18804331
- [Result] Heck JE, Stucker I, Allwright S, Gritz ER, Haglund M, Healton CG, Kralikova E, Sanchez Del Mazo S, Tamang E, Dresler CM, Hashibe M. Home and workplace smoking bans in Italy, Ireland, Sweden, France and the Czech Republic. Eur Respir J. 2010 May;35(5):969-79. doi: 10.1183/09031936.00066809. Epub 2009 Nov 19. PMID 19926747
- [Result] Hill SC, Liang L. Smoking in the home and children's health. Tob Control. 2008 Feb;17(1):32-7. doi: 10.1136/tc.2007.020990. PMID 18218804
- [Result] Ho SY, Wang MP, Lo WS, Mak KK, Lai HK, Thomas GN, Lam TH. Comprehensive smoke-free legislation and displacement of smoking into the homes of young children in Hong Kong. Tob Control. 2010 Apr;19(2):129-33. doi: 10.1136/tc.2009.032003. PMID 20378586
- [Result] Hollis JF, McAfee TA, Fellows JL, Zbikowski SM, Stark M, Riedlinger K. The effectiveness and cost effectiveness of telephone counselling and the nicotine patch in a state tobacco quitline. Tob Control. 2007 Dec;16 Suppl 1(Suppl 1):i53-9. doi: 10.1136/tc.2006.019794. PMID 18048633
- [Result] Hovell MF, Meltzer SB, Wahlgren DR, Matt GE, Hofstetter CR, Jones JA, Meltzer EO, Bernert JT, Pirkle JL. Asthma management and environmental tobacco smoke exposure reduction in Latino children: a controlled trial. Pediatrics. 2002 Nov;110(5):946-56. doi: 10.1542/peds.110.5.946. PMID 12415035
- [Result] Hovell MF, Zakarian JM, Matt GE, Hofstetter CR, Bernert JT, Pirkle J. Effect of counselling mothers on their children's exposure to environmental tobacco smoke: randomised controlled trial. BMJ. 2000 Aug 5;321(7257):337-42. doi: 10.1136/bmj.321.7257.337. PMID 10926589
- [Result] Hovell MF, Zakarian JM, Matt GE, Liles S, Jones JA, Hofstetter CR, Larson SN, Benowitz NL. Counseling to reduce children's secondhand smoke exposure and help parents quit smoking: a controlled trial. Nicotine Tob Res. 2009 Dec;11(12):1383-94. doi: 10.1093/ntr/ntp148. Epub 2009 Oct 29. PMID 19875762
- [Result] Hoving EF, Mudde AN, de Vries H. Predictors of smoking relapse in a sample of Dutch adult smokers; the roles of gender and action plans. Addict Behav. 2006 Jul;31(7):1177-89. doi: 10.1016/j.addbeh.2005.09.002. Epub 2005 Oct 19. PMID 16242246
- [Result] Huang HL, Yen YY, Lin PL, Chiu CH, Hsu CC, Chen T, Hu CY, Lin YY, Lee CH, Chen FL. Household secondhand smoke exposure of elementary schoolchildren in Southern Taiwan and factors associated with their confidence in avoiding exposure: a cross-sectional study. BMC Public Health. 2012 Jan 17;12:40. doi: 10.1186/1471-2458-12-40. PMID 22251625
- [Result] Hugg TT, Jaakkola MS, Ruotsalainen RO, Pushkarev VJ, Jaakkola JJ. Parental smoking behaviour and effects of tobacco smoke on children's health in Finland and Russia. Eur J Public Health. 2008 Feb;18(1):55-62. doi: 10.1093/eurpub/ckm053. Epub 2007 Jun 14. PMID 17569700
- [Result] Hughes SC, Corcos IA, Hofstetter CR, Hovell MF, Irvin VL. Longitudinal study of household smoking ban adoption among Korean Americans. Am J Prev Med. 2009 Nov;37(5):437-40. doi: 10.1016/j.amepre.2009.06.015. PMID 19840699
- [Result] Hyland A, Higbee C, Travers MJ, Van Deusen A, Bansal-Travers M, King B, Cummings KM. Smoke-free homes and smoking cessation and relapse in a longitudinal population of adults. Nicotine Tob Res. 2009 Jun;11(6):614-8. doi: 10.1093/ntr/ntp022. Epub 2009 Apr 3. PMID 19346505
- [Result] Lampert T. Smoking and passive smoking exposure in young people: results of the German Health Interview and Examination Survey for Children and Adolescents (KiGGS). Dtsch Arztebl Int. 2008 Apr;105(15):265-71. doi: 10.3238/arztebl.2008.0265. Epub 2008 Apr 11. PMID 19629230
- [Result] Li MF, Wang RH. Factors related to avoidance of environmental tobacco smoke among adolescents in southern Taiwan. J Nurs Res. 2006 Jun;14(2):103-12. doi: 10.1097/01.jnr.0000387568.41941.f0. PMID 16741860
- [Result] Martinelli AM. Development and validation of the avoidance of environmental tobacco smoke scale. J Nurs Meas. 1998 Summer;6(1):75-86. PMID 9769612
- [Result] Matt GE, Quintana PJ, Hovell MF, Bernert JT, Song S, Novianti N, Juarez T, Floro J, Gehrman C, Garcia M, Larson S. Households contaminated by environmental tobacco smoke: sources of infant exposures. Tob Control. 2004 Mar;13(1):29-37. doi: 10.1136/tc.2003.003889. PMID 14985592
- [Result] Mills AL, Messer K, Gilpin EA, Pierce JP. The effect of smoke-free homes on adult smoking behavior: a review. Nicotine Tob Res. 2009 Oct;11(10):1131-41. doi: 10.1093/ntr/ntp122. Epub 2009 Jul 24. PMID 19633273
- [Result] Mills LM, Semple SE, Wilson IS, MacCalman L, Amos A, Ritchie D, O'Donnell R, Shaw A, Turner SW. Factors influencing exposure to secondhand smoke in preschool children living with smoking mothers. Nicotine Tob Res. 2012 Dec;14(12):1435-44. doi: 10.1093/ntr/nts074. Epub 2012 Mar 15. PMID 22422926
- [Result] Moore GF, Currie D, Gilmore G, Holliday JC, Moore L. Socioeconomic inequalities in childhood exposure to secondhand smoke before and after smoke-free legislation in three UK countries. J Public Health (Oxf). 2012 Dec;34(4):599-608. doi: 10.1093/pubmed/fds025. Epub 2012 Mar 23. PMID 22448041
- [Result] Nattala P, Leung KS, Nagarajaiah, Murthy P. Family member involvement in relapse prevention improves alcohol dependence outcomes: a prospective study at an addiction treatment facility in India. J Stud Alcohol Drugs. 2010 Jul;71(4):581-7. doi: 10.15288/jsad.2010.71.581. PMID 20553667
- [Result] Nierkens V, Stronks K, van Oel CJ, de Vries H. Beliefs of Turkish and Moroccan immigrants in The Netherlands about smoking cessation: implications for prevention. Health Educ Res. 2005 Dec;20(6):622-34. doi: 10.1093/her/cyh026. Epub 2005 Mar 21. PMID 15781443
- [Result] Phillips R, Amos A, Ritchie D, Cunningham-Burley S, Martin C. Smoking in the home after the smoke-free legislation in Scotland: qualitative study. BMJ. 2007 Sep 15;335(7619):553. doi: 10.1136/bmj.39301.497593.55. Epub 2007 Sep 9. PMID 17827488
- [Result] Roseby R, Waters E, Polnay A, Campbell R, Webster P, Spencer N. Family and carer smoking control programmes for reducing children's exposure to environmental tobacco smoke. Cochrane Database Syst Rev. 2003;(3):CD001746. doi: 10.1002/14651858.CD001746. PMID 12917911
- [Result] Prochaska JO, Velicer WF, Redding C, Rossi JS, Goldstein M, DePue J, Greene GW, Rossi SR, Sun X, Fava JL, Laforge R, Rakowski W, Plummer BA. Stage-based expert systems to guide a population of primary care patients to quit smoking, eat healthier, prevent skin cancer, and receive regular mammograms. Prev Med. 2005 Aug;41(2):406-16. doi: 10.1016/j.ypmed.2004.09.050. PMID 15896835
- [Result] Robinson J, Kirkcaldy AJ. Disadvantaged mothers, young children and smoking in the home: mothers' use of space within their homes. Health Place. 2007 Dec;13(4):894-903. doi: 10.1016/j.healthplace.2007.03.001. Epub 2007 Mar 21. PMID 17499542
- [Result] Robinson J, Kirkcaldy AJ. 'You think that I'm smoking and they're not': why mothers still smoke in the home. Soc Sci Med. 2007 Aug;65(4):641-52. doi: 10.1016/j.socscimed.2007.03.048. Epub 2007 May 7. PMID 17482738
- [Result] Robinson J, Kirkcaldy AJ. 'Imagine all that smoke in their lungs': parents' perceptions of young children's tolerance of tobacco smoke. Health Educ Res. 2009 Feb;24(1):11-21. doi: 10.1093/her/cym080. Epub 2007 Dec 20. PMID 18156146
- [Result] Rosen LJ, Ben Noach M. Systematic reviews on tobacco control from Cochrane and the Community Guide: different methods, similar findings. J Clin Epidemiol. 2010 Jun;63(6):596-606. doi: 10.1016/j.jclinepi.2009.09.010. Epub 2010 Jan 13. PMID 20056382
- [Result] Rosen LJ, Noach MB, Winickoff JP, Hovell MF. Parental smoking cessation to protect young children: a systematic review and meta-analysis. Pediatrics. 2012 Jan;129(1):141-52. doi: 10.1542/peds.2010-3209. Epub 2011 Dec 26. PMID 22201152
- [Result] Poole-Di Salvo E, Liu YH, Brenner S, Weitzman M. Adult household smoking is associated with increased child emotional and behavioral problems. J Dev Behav Pediatr. 2010 Feb-Mar;31(2):107-15. doi: 10.1097/DBP.0b013e3181cdaad6. PMID 20110826
- [Result] Schumann A, John U, Ulbricht S, Ruge J, Bischof G, Meyer C. Computer-generated tailored feedback letters for smoking cessation: theoretical and empirical variability of tailoring. Int J Med Inform. 2008 Nov;77(11):715-22. doi: 10.1016/j.ijmedinf.2008.03.001. Epub 2008 Apr 15. PMID 18417417
- [Result] Tanner-Smith EE, Wilson SJ, Lipsey MW. The comparative effectiveness of outpatient treatment for adolescent substance abuse: a meta-analysis. J Subst Abuse Treat. 2013 Feb;44(2):145-58. doi: 10.1016/j.jsat.2012.05.006. Epub 2012 Jul 2. PMID 22763198
- [Result] Tyc VL, Hovell MF, Winickoff J. Reducing secondhand smoke exposure among children and adolescents: emerging issues for intervening with medically at-risk youth. J Pediatr Psychol. 2008 Mar;33(2):145-55. doi: 10.1093/jpepsy/jsm135. Epub 2008 Jan 11. PMID 18192298
- [Result] Tyc VL, Huang Q, Nicholson J, Schultz B, Hovell MF, Lensing S, Vukadinovich C, Hudson MM, Zhang H. Intervention to reduce secondhand smoke exposure among children with cancer: a controlled trial. Psychooncology. 2013 May;22(5):1104-11. doi: 10.1002/pon.3117. Epub 2012 Jun 8. PMID 22684982
- [Result] Wagener TL, Gregor KL, Busch AM, McQuaid EL, Borrelli B. Risk perception in smokers with children with asthma. J Consult Clin Psychol. 2010 Dec;78(6):980-5. doi: 10.1037/a0021094. PMID 21114346
- [Result] Wamboldt FS, Balkissoon RC, Rankin AE, Szefler SJ, Hammond SK, Glasgow RE, Dickinson WP. Correlates of household smoking bans in low-income families of children with and without asthma. Fam Process. 2008 Mar;47(1):81-94. doi: 10.1111/j.1545-5300.2008.00240.x. PMID 18411831
- [Result] Wang WL, Herting JR, Tung YY. Adolescents' avoidance of secondhand smoke exposure: model testing. West J Nurs Res. 2008 Nov;30(7):836-51. doi: 10.1177/0193945908319251. Epub 2008 May 30. PMID 18515750
- [Result] Wilkinson AV, Shete S, Prokhorov AV. The moderating role of parental smoking on their children's attitudes toward smoking among a predominantly minority sample: a cross-sectional analysis. Subst Abuse Treat Prev Policy. 2008 Jul 14;3:18. doi: 10.1186/1747-597X-3-18. PMID 18625061
- [Result] Wilson SR, Farber HJ, Knowles SB, Lavori PW. A randomized trial of parental behavioral counseling and cotinine feedback for lowering environmental tobacco smoke exposure in children with asthma: results of the LET'S Manage Asthma trial. Chest. 2011 Mar;139(3):581-590. doi: 10.1378/chest.10-0772. Epub 2010 Sep 23. PMID 20864611
- [Result] Winickoff JP, Friebely J, Tanski SE, Sherrod C, Matt GE, Hovell MF, McMillen RC. Beliefs about the health effects of "thirdhand" smoke and home smoking bans. Pediatrics. 2009 Jan;123(1):e74-9. doi: 10.1542/peds.2008-2184. PMID 19117850
- [Result] Woods SE, Springett J, Porcellato L, Dugdill L. 'Stop it, it's bad for you and me': experiences of and views on passive smoking among primary-school children in Liverpool. Health Educ Res. 2005 Dec;20(6):645-55. doi: 10.1093/her/cyh027. Epub 2005 Apr 13. PMID 15829496
- [Result] Wu D, Ma GX, Zhou K, Zhou D, Liu A, Poon AN. The effect of a culturally tailored smoking cessation for Chinese American smokers. Nicotine Tob Res. 2009 Dec;11(12):1448-57. doi: 10.1093/ntr/ntp159. Epub 2009 Nov 13. PMID 19915080
- [Result] Yilmaz G, Karacan C, Yoney A, Yilmaz T. Brief intervention on maternal smoking: a randomized controlled trial. Child Care Health Dev. 2006 Jan;32(1):73-9. doi: 10.1111/j.1365-2214.2006.00570.x. PMID 16398793
- [Result] Young JM, Girgis S, Bruce TA, Hobbs M, Ward JE. Acceptability and effectiveness of opportunistic referral of smokers to telephone cessation advice from a nurse: a randomised trial in Australian general practice. BMC Fam Pract. 2008 Feb 28;9:16. doi: 10.1186/1471-2296-9-16. PMID 18304363
- [Result] Yousey Y. Family attitudes about tobacco smoke exposure of young children at home. MCN Am J Matern Child Nurs. 2007 May-Jun;32(3):178-83. doi: 10.1097/01.NMC.0000269568.17432.72. PMID 17479055
- [Result] Zakarian JM, Hovell MF, Sandweiss RD, Hofstetter CR, Matt GE, Bernert JT, Pirkle J, Hammond SK. Behavioral counseling for reducing children's ETS exposure: implementation in community clinics. Nicotine Tob Res. 2004 Dec;6(6):1061-74. doi: 10.1080/1462220412331324820. PMID 15801580